CLINICAL TRIAL: NCT01221441
Title: A Phase II Study to Determine the Efficacy and Safety of Allogeneic Human Chondrocytes Expressing TGF-β1 (TissueGene-C) in Patients With Grade 3 Chronic Degenerative Joint Disease of the Knee
Brief Title: Study of TG-C in Patients With Grade 3 Degenerative Joint Disease of the Knee
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kolon TissueGene, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TGC09201
Record Dates: First submitted 2010-10-13; First posted 2010-10-15 (Estimated); Results first posted 2016-02-15 (Estimated); Last update posted 2016-02-15 (Estimated); Status verified 2016-01

CONDITIONS: Osteoarthritis, Knee
Keywords: Cartilage; Knee; Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TissueGene-C (Experimental): TissueGene-C at 3 x 10e7 cells per injection (intraarticular)
  Interventions: Biological: TissueGene-C
- Placebo Control (Placebo Comparator): Normal Saline injection
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: TissueGene-C — Single intraarticular injection at 3 x 10e7 cells
  Other Names: TG-C
  Arms: TissueGene-C
Drug: Normal Saline — Single intraarticular injection of normal saline as a placebo control
  Other Names: 0.9% Saline
  Arms: Placebo Control

SUMMARY:
The purpose of this study is to see if we can safely regenerate cartilage without invasive surgery using a biologic product called TissueGene-C.

DETAILED DESCRIPTION:
Protocol TGC09201 is a multi-center, double-blind, placebo-controlled, randomized study. A total of one hundred (100) adults with grade 3 chronic degenerative joint disease (DJD) of the knee joint (as determined by radiographic examination) will be enrolled into the study. TissueGene-C will be administered intra-articularly once via x-ray guidance. TissueGene-C will be administered at a dose of 3 x 10e7 cells. Patients receiving control treatment will receive a single normal saline injection.

The objectives of this study are to:

1. Evaluate the efficacy of TissueGene-C with regard to knee functionality and symptoms of knee osteoarthritis including pain.
2. Evaluate the safety of administration of a single intra-articular dose of TissueGene-C as evidenced by observation of the injection site for irritation or other abnormalities, the incidence and severity of adverse events, and the changes in physical examination findings and laboratory tests, including immune analyses.
3. Evaluate the incidence and dose of analgesia and/or anti-inflammatory medication.
4. Evaluate the regeneration of hyaline cartilage as determined by 3T magnetic resonance imaging (MRI).
5. Evaluate distribution of hChonJb#7 cells out of the injection site.
6. Evaluate the efficacy of TissueGene-C by evaluating the need for total knee arthroplasty after treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female subject
2. Age 18 to 70 years
3. In general good health as evidenced by physical examination, normal hematology, serum chemistry, and urinalysis screening laboratory results, and a negative history of significant organ system disorders. All laboratory values must be within 20% of normal ranges.

   1. Body Mass Index (BMI) should be between '18.5 - 45.5'. The applied scale is the same for both men and women.
   2. Blood Pressure measurements - Systolic Blood Pressure should be between 90-160mm. Hg, and Diastolic Blood Pressure between 50-90mm.Hg,
4. Patients with Grade 3 chronic osteoarthritis of the knee as determined by the Radiographic Criteria of Kellgren and Lawrence.
5. Symptom of pain for more than four (4) consecutive months and intensity of ≥ 40 and ≤ 90 on the 100-mm scale.
6. Patients should be cleared to use protocol specified equipment: 3T MRI.
7. Patients providing written informed consent after the nature of the study is fully explained and understood by the patient.

Exclusion Criteria:

1. Age 71 or older
2. Patients with abnormal hematology, serum chemistry, or urinalysis screening laboratory results.
3. Patients taking non-steroidal anti-inflammatory medications within 14 days of baseline visit unless washed out as per section 3.6.4 above.
4. Patients taking steroidal anti-inflammatory medications within 2 months of baseline visit.
5. Patients with a recent (within 1 year) history of drug abuse and/or a positive urine drug test at the time of screening.
6. Patients receiving injections to the treated knee within 2 months prior to study entry
7. Patients who are contraindicated for 3T MRI.
8. Patients who are pregnant or currently breast-feeding children.
9. Patients with systemic, rheumatic or inflammatory disease of the knee or chondrocalcinosis, hemochromatosis, inflammatory arthritis, necrosis of the femoral condyle, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, infectious arthritis, Charcot's knee joint, villonodular synovitis, synovial chondromatosis, and/or history of inflammatory arthropathy.
10. Patients with ongoing infectious disease, including HIV and hepatitis B or C.
11. Patients with clinically significant cardiovascular, renal, hepatic, endocrine disease, cancer, or Type I diabetes.
12. Patients participating in a study of an experimental drug or medical device within 30 days of study entry.
13. Patients that will be unable to comply with the requisite study follow-up and are not able to complete all of the follow-up office visits and 3T MRI exams.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2011-05; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Mont, MD, Principal Investigator — Sinai Hospital of Baltimore; David W Romness, MD, Principal Investigator — Commonwealth Orthopedics, Virginia Hospital Center
Locations (5):
- United States (5):
  - Advent Clinical Research, Pinellas Park, Florida
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - Rothman Institute, Philadelphia, Pennsylvania
  - University Orthopedics, State College, Pennsylvania
  - Commonwealth Orthopedics, Arlington, Virginia

REFERENCES:
- [Derived] Guermazi A, Kalsi G, Niu J, Crema MD, Copeland RO, Orlando A, Noh MJ, Roemer FW. Structural effects of intra-articular TGF-beta1 in moderate to advanced knee osteoarthritis: MRI-based assessment in a randomized controlled trial. BMC Musculoskelet Disord. 2017 Nov 16;18(1):461. doi: 10.1186/s12891-017-1830-8. PMID 29145839
- [Derived] Cherian JJ, Parvizi J, Bramlet D, Lee KH, Romness DW, Mont MA. Preliminary results of a phase II randomized study to determine the efficacy and safety of genetically engineered allogeneic human chondrocytes expressing TGF-beta1 in patients with grade 3 chronic degenerative joint disease of the knee. Osteoarthritis Cartilage. 2015 Dec;23(12):2109-2118. doi: 10.1016/j.joca.2015.06.019. Epub 2015 Jul 16. PMID 26188189

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TissueGene-C | Placebo Control
Started | 67 | 35
Completed | 45 | 23
Not Completed | 22 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TissueGene-C | Placebo Control | Total
Number analyzed (Participants) | 67 | 35 | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 20 | 59
  >=65 years | 28 | 15 | 43
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.7 (7.89) | 56.5 (8.62) | 56.6 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 21 | 64
  Male | 24 | 14 | 38
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian/White | 53 | 29 | 82
  Black | 12 | 4 | 16
  Hispanic | 2 | 2 | 4
Region of Enrollment [Number; unit: participants]
  United States | 67 | 35 | 102
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.6 (5.87) | 29.6 (5.62) | 29.6 (5.70)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation Score at 1 Year
Description: Symptoms, pain and function of the knee joint determined and scored using the International Knee Documentation Committee (IKDC) Subjective Knee Evaluation (Total Score, range 0-100 with higher scores better). Linear mixed model used for analysis.
Time Frame: 1 Year
Population: Patients with available baseline IKDC scores
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 38 | 20
scores on a scale | 23.3 [17.3 to 29.3] | 9.9 [1.7 to 18.1]
Statistical Analysis 1: Comparison: TissueGene-C vs Placebo Control; The primary efficacy evaluation based on IKDC and the VAS were tested at week 52 evaluated 100 mm VAS with the following superiority hypothesis: HO: μTG = μPC vs. HA: μTG ≠ μPC, where μTG and μPC are the mean change from baseline in IKDC or VAS scores at week 52 for patients in the TG-C and placebo control groups, respectively. If the null hypotheses for both the IKDC and the VAS are rejected, it the clinical effect of TG-C is concluded to be superior to that of the control; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Denominator degrees of freedom were adjusted using the Kenward-Roger's method

2. Primary Outcome: Change From Baseline in Visual Analog Scale (VAS) Score at 1 Year
Description: Reduction in pain as measured by a 100 mm visual analog scale (0= no pain; 100 = extreme pain) from Baseline to 1 Year. Linear mixed model used for analysis.
Time Frame: 1 Year
Population: Patients with available baseline and 1 year VAS score
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 49 | 24
units on a scale | -39.7 [-46.7 to -32.7] | -24.3 [-34.1 to -14.5]
Statistical Analysis 1: Comparison: TissueGene-C vs Placebo Control; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Denominator degrees of freedom were adjusted using the Kenward-Roger's method

3. Secondary Outcome: Change From Baseline in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 2 Years
Description: Symptoms, pain and functionality of the knee joint as determined by Total Score of the Knee Injury and Osteoarthritis Outcome Score (KOOS) (Range 0-100 with higher scores indicating healthier outcomes). Linear mixed model used for analysis.
Time Frame: 2 Years
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 45 | 23
scores on a scale | 10.0 [6.0 to 13.9] | 10.5 [5.0 to 16.0]
Statistical Analysis 1: Comparison: TissueGene-C vs Placebo Control; The efficacy evaluation at week 104 evaluated KOOS with the following superiority hypothesis: HO: μTG = μPC vs. HA: μTG ≠ μPC, where μTG and μPC are the mean change from baseline in KOOS scores at week 104 for patients in the TG-C and placebo control groups, respectively. If the null hypotheses for KOOS is rejected, it the clinical effect of TG-C is concluded to be superior to that of the control; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Denominator degrees of freedom were adjusted using the Kenward-Roger's method

4. Secondary Outcome: Change From Baseline in Articular Cartilage Damage in the Knee as Determined by the Lysholm Knee Score at 2 Years
Description: Measurement to assess outcomes of various chondral disorders of the knee determined by the Lysholm Knee Scale (Range 0-100 with higher scores better). Linear mixed model used for analysis.
Time Frame: 2 Years
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 45 | 23
scores on a scale | 20.1 [14.8 to 25.5] | 11.4 [4.1 to 18.8]
Statistical Analysis 1: Comparison: TissueGene-C vs Placebo Control; The efficacy evaluation at week 104 evaluated Lysholm score with the following superiority hypothesis: HO: μTG = μPC vs. HA: μTG ≠ μPC, where μTG and μPC are the mean change from baseline in KOOS scores at week 104 for patients in the TG-C and placebo control groups, respectively. If the null hypotheses for Lysholm score is rejected, it the clinical effect of TG-C is concluded to be superior to that of the control; Test type: Superiority or Other; p < 0.01, Mixed Models Analysis; Denominator degrees of freedom were adjusted using the Kenward-Roger's method

5. Secondary Outcome: Comparative Evaluation of Knee Magnetic Resonance Images (MRIs) From Baseline to 1 Year
Description: Comparison of pre-procedure 3T MRI scans to those obtained at months 12 following dose administration by an independent radiographic reviewer. Evaluations will be scored using Whole Organ Magnetic Resonance imaging Score (WORMS) Cartilage Morphology Subscore (Range 0-6, with higher scores being worse)
Time Frame: 1 Year
Population: Patients with available baseline and 1-year MRIs
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 32 | 22
scores on a scale | 0.03 [-1.22 to 1.29] | -0.49 [-2.07 to 1.08]

6. Secondary Outcome: Change in Pain Severity From Baseline to 2 Years as Assessed by Questionnaire
Description: Change in pain severity (on a scale from 1 to 4) from baseline to 2 years as measured by a questionnaire (lower scores better)
Time Frame: 2 Years
Population: Patients that completed 2 year follow-up
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 33 | 18
scores on a scale | -0.87 (0.844) | -0.30 (1.031)

7. Secondary Outcome: Number of Participants With Change in Pain Severity Measured by Incidence and Dose of Analgesia
Description: The number of participants that had a change in pain severity as measured by the incidence and dose of analgesic medications
Time Frame: 2 Years
Population: Patients taking at least one analgesia medication
Measure: Number; unit: participants
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 67 | 35
participants | 37 | 20

8. Secondary Outcome: Change From Baseline in Knee Function as Determined by the Lower Extremity Functional Scale at 2 Years
Description: Assessment of knee function as determined by the Lower Extremity Functional Scale (LEFS); change from baseline to 2 years (Range 0-80 with higher scores signifying lower difficulty in performing knee functions)
Time Frame: 2 Years
Population: Patients that completed 2-year follow-up
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 45 | 23
scores on a scale | 16.7 [11.9 to 21.5] | 13.8 [7.1 to 20.4]

9. Secondary Outcome: The Incidence of Total Knee Arthroplasty
Description: Quantification of the incidence of total knee arthroplasty of the treated knee subsequent to treatment with TissueGene-C
Time Frame: 2 Years
Population: All patients that participated in the study
Measure: Number; unit: participants
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 67 | 35
participants | 1 | 1

10. Secondary Outcome: The Number of Patients Experiencing Injection Site Reactions Related to Treatment
Description: The number of patients with observations of the administration site deemed related to treatment with either active or placebo, including arthralgia, swelling, irritation, pain, stiffness or abnormalities
Time Frame: 2 Years
Population: All participants receiving placebo or active treatment
Measure: Number; unit: participants
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 67 | 35
participants | 35 | 5

11. Secondary Outcome: The Incidence and Severity of Adverse Events in Treated Patients
Description: The incidence and severity of adverse events assessed through 104 weeks (2 years) after dose administration
Time Frame: 2 Years
Population: All patients receiving treatment with either active or placebo
Measure: Number; unit: participants
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 67 | 35
participants
  Mild | 12 | 7
  Moderate | 41 | 18
  Severe | 8 | 4

12. Secondary Outcome: Number of Participants With Adverse Events Due to Clinically Significant Changes in Hematology and Urinalysis Tests
Description: The number of participants with changes in clinical hematology, chemistry, and urinalysis test results through 2 years that were considered Adverse Events
Time Frame: 2 Years
Population: All patients
Measure: Number; unit: participants
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 67 | 35
participants | 17 | 5

13. Secondary Outcome: Change in SF-36 General Health Assessment Questionnaire (Overall Score) From Baseline to 2 Years
Description: Overall assessment of general health as determined by scoring use an SF-36 Questionnaire (Range 0-100 with higher scores better - indicating less disability)
Time Frame: 2 Years
Population: Patients with completed SF-36 questionnaire at 104 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: scores on a scale
Arm/Group | TissueGene-C | Placebo Control
Number analyzed (Participants) | 45 | 22
scores on a scale | 7.6 [4.4 to 10.8] | 6.7 [2.2 to 11.2]

ADVERSE EVENTS:
Arm/Group | TissueGene-C | Placebo Control
Serious Adverse Events (participants affected / at risk) | 7/67 | 4/35
Other Adverse Events (participants affected / at risk) | 45/67 | 8/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TissueGene-C (N=67) | Placebo Control (N=35)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Radius Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Total Knee Arthroplasty (Surgical and medical procedures) | 2 (2) | 1 (1)
Hiatal hernia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Invertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Microdiscectomy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Prostatectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Column Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal Fusion Surgery (Surgical and medical procedures) | 1 (1) | 1 (1)
Spinal Laminectomy (Surgical and medical procedures) | 1 (1) | 1 (1)
Invertebral Disc Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Lumbar Degenerative Disc Disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TissueGene-C (N=67) | Placebo Control (N=35)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Feeling Cold (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
C-reactive Protein Increased (Investigations) | 1 (1) | 0 (0)
Eosinophil Count Increased (Investigations) | 1 (1) | 0 (0)
Interleukin Level Increased (Investigations) | 5 (5) | 1 (1)
Red Blood Cell Sedimentation Increased (Investigations) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (15) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 19 (19) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint Effusions (Musculoskeletal and connective tissue disorders) | 13 (13) | 2 (2)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weight Bearing Difficulty (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin Warm (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Increased White Blood Cells/Neutrophils (Investigations) | 1 (1) | 0 (0)
Right Knee Swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No